CLINICAL TRIAL: NCT05038540
Title: Evaluation of the Effect of Virtual Reality Glasses Used During Scaling and Root Planing on Dental Anxiety Control
Brief Title: The Effect of Virtual Reality Glasses on Dental Anxiety Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ezgi Gürbüz, Assistant Professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00
Record Dates: First submitted 2021-09-03; First posted 2021-09-09 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Periodontitis; Dental Anxiety; Dental Fear; Gingivitis; Calculus, Dental
MeSH Terms: conditions — Periodontitis; Gingivitis; Dental Calculus | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality application (Experimental): Application of virtual reality glasses during scaling and root planning to a quadrant.
  Interventions: Procedure: Scaling and root planing
- No application (Active Comparator): No application of virtual reality glasses during scaling and root planning to a quadrant.
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Procedure: Scaling and root planing — Phase 1 periodontal therapy

SUMMARY:
In this clinical study, it was aimed to evaluate whether there is a decrease in patient anxiety by applying virtual reality glasses, which are the product of new technology, during scaling and root planing treatment.

Patients who required scaling and root planing treatment and also scored 9 or above according to the Dental Anxiety Scale were included in our study. Scaling and root planing was performed in a randomly selected intraoral quadrant of the patients, in the same way, with or without the use of virtual reality glasses. In the virtual reality glasses application, a video consisting of images of nature landscapes developed for patient rehabilitation was projected onto the screen in front of the patient's eyes. The Dental Anxiety Scale was reapplied after the completion of the treatment.

In the intraoral quadrant where virtual reality glasses were used, it is expected that lower Corah Dental Anxiety Scale scores may be obtained after the treatment is completed, compared to the intraoral quadrant where the treatment is performed without glasses, thus reducing anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being systemically healthy
* Needing treatment in at least two quadrants of the mouth
* At least five teeth in each quadrant and at least one region with a terminal pocket depth ≥4 mm
* Having a score of 9 or higher on the dental anxiety scale

Exclusion Criteria:

* Having a history of seizures or a convulsive disorder
* Balance disorders such as nystagmus, vertigo
* Use of psychotropic drugs
* Getting treatment for anxiety
* Presence of dermatological lesions on the face and especially around the eyes
* The presence of a lesion in the eye that will prevent the use of virtual reality glasses

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Lower Corah Dental Anxiety Scale scores in virtual reality application group | Baseline
  It is expected that lower Corah Dental Anxiety Scale scores may be obtained after the treatment is completed, compared to the intraoral quadrant where the treatment is performed without glasses, thus reducing anxiety.
Lower blood pressure and heart rate values in virtual reality application group | Baseline
  It is expected that lower blood pressure and heart rate values will be obtained during and after treatment in the intraoral quadrant, where glasses are used, compared to the control quadrant.

SECONDARY OUTCOMES:
Patients' feedback | Baseline, 1st month
  It is expected that positive feedback will be received by evaluating the patients' feelings. about the glasses application with the Visual Analog Scale applied after the treatment is completed.
Dentist's feedback | Baseline
  After the treatment, it is expected that the use of glasses in patients with anxiety will be evaluated as a viable method by taking the opinions of the physicians regarding the application.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)